CLINICAL TRIAL: NCT00714766
Title: Heat Stress and Volume Administration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Niels Secher, Professor, Righospitale
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Heat stress RH08
Record Dates: First submitted 2008-07-10; First posted 2008-07-14 (Estimated); Last update posted 2009-02-16 (Estimated); Status verified 2009-02

CONDITIONS: Syncope
MeSH Terms: conditions — Syncope

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- A (Experimental)
  Interventions: Procedure: Intravascular volume administration

INTERVENTIONS:
Procedure: Intravascular volume administration — Infusion of colloid to reestablish CVP under heat stress

SUMMARY:
Heat stress reduces the central blood volume and causes orthostatic intolerance. The hypothesis is that infusion of volume may reduce effects of orthostatic stress during heat stress.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 < 40

Exclusion Criteria:

* Abnormal medical history

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2008-07; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Cardiac filling pressure in relation to cardiac SV | with varying degress of lower body negative pressures

CONTACTS AND LOCATIONS:
Overall Officials: Niels Secher, MD, PhD, Study Director — Rigshospitalet, Denmark
Locations (1):
- Dept of anesthesiology 2041, Copenhagen, Denmark